CLINICAL TRIAL: NCT07342218
Title: Pilot Trial of Digital Substance Use Disorder Interventions to Prevent Post-release Substance Use Disorder Relapse in Offenders in Correctional Service of Canada Custody
Brief Title: Correctional Service of Canada Pilot Trial of Digital Substance Use Disorder Interventions (PROCESS)
Acronym: PROCESS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Correctional Service of Canada (Other Government)
Responsible Party: Principal Investigator, James MacKillop, Director, Peter Boris Centre for Addiction Research; Director, Michael G. DeGroote Centre for Medicinal Cannabis Research, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18879; Memorandum of Understanding (Other: Correctional Service of Canada)
Record Dates: First submitted 2025-12-08; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-11

CONDITIONS: Substance Use Disorder (SUD)
Keywords: incarceration; federal offender; substance use disorder; cognitive behavioural therapy; mindfulness; digital treatment; substance use treatment; pilot trial
MeSH Terms: conditions — Substance-Related Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computer-Based Training for Cognitive Behavioural Therapy (Experimental): Participants will complete a 7-module digital treatment intervention for substance use, using cognitive behavioural therapy practices.
  Interventions: Other: Computer-Based Training for Cognitive Behavioural Therapy (CBT4CBT)
- Breaking Free Online (Experimental): Participants will complete a 6-module digital treatment intervention for substance use, using cognitive behavioural therapy and mindfulness techniques.
  Interventions: Other: Breaking Free Online (BFO)

INTERVENTIONS:
Other: Breaking Free Online (BFO) — BFO is a digital intervention for substance use problems and commonly co-occurring disorders, such as depression and anxiety. Its structure is based on cognitive behavioural therapy (CBT) and mindfulness techniques. It is self-directed by the individual and can be done on a smartphone, tablet, or online. BFO provides techniques for cognitive restructuring (i.e., reshaping how we view certain situations) and managing and planning for high-risk situations (e.g., minimizing relapse in the face of certain triggers).
  Arms: Breaking Free Online
Other: Computer-Based Training for Cognitive Behavioural Therapy (CBT4CBT) — CBT4CBT is a digital intervention used for substance use problems through the application of CBT techniques. The program involves various video modules, educational games, quizzes, interactive videos, and more. The modules are self-paced and can be done online. Modules will focus on teaching users core skills to avoid substance use and ways of effectively communicating. It discusses various situations where potential triggers could arise, and homework done afterwards allows the user to identify their own personal triggers and individualize how they can minimize these risks.
  Arms: Computer-Based Training for Cognitive Behavioural Therapy

SUMMARY:
Problems with substance use are common in prisoners. Since most substances are still illegal in Canada, substance use problems can increase the risk for re-incarceration. Although research suggests that treatment may reduce these risks, they are still rarely used in correctional settings. This pilot study will examine the feasibility and usefulness of two digital treatments for substance use problems in individuals recently released from prison. The investigators will compare engagement across both treatments over a 6-month period, and assess the rates of substance use relapse and re-incarceration.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have previously served custodial services in the Correctional Services of Canada (csc).
* Individuals who have a history of substance use problems (i.e., determined by them not being allowed to use substances as part their parole terms)
* Individuals who current reside in a Community Correctional Centre or Community-Based Residential Facility
* Individuals between 18-55 years old

Exclusion Criteria:

- Individuals who have never served a custodial sentence with the CSC

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Digital Treatment Interventions | End of enrollment (~6 months)
  Number of enrolled pilot trial participants, overall and by intervention.
Overall Substance Use Treatment Engagement | End of enrollment (~6 months)
  The number and percentage of modules, and homework modules, completed.
Perceived Treatment Utility | End of enrollment (~6 months)
  Mean module and overall treatment rating using a 4-question "Module Utility" scale created by the research team. This is an 11-point Likert scale (0-10) rating the importance, relevance, usefulness, and likeliness to recommend treatment, with higher scores indicating better utility.
Efficacy of Treatment Module Content | End of enrollment (~6 months)
  Treatment modules include quizzes with several true or false questions (5-10 questions per module) that assess individuals' understanding of the content learned. Overall performance on intervention quizzes in treatment modules will be examined using the total number of questions answered correctly, with higher scores indicating a better understanding of the treatment modules.
Efficacy of Digital Treatment Interventions for Substance Use | Study follow-up (~3 months post-treatment completion)
  Substance use relapse documented by the CSC staff.
Efficacy of Digital Treatment Interventions for Recidivism | Study follow-up (~3 months post-treatment completion)
  Institutional readmission documented by the CSC staff.

SECONDARY OUTCOMES:
Between-Intervention Feasibility Outcomes | End of enrollment (~6 months)
  Comparing treatment utility ratings on the 4-question "Module Utility" questionnaire between interventions.
Between-Intervention Efficacy Outcomes for Substance Use | Study follow-up (~3 months post-treatment completion)
  Comparing substance use relapse as documented by CSC staff between treatment groups.
Between-Intervention Efficacy Outcomes for Recidivism | Study follow-up (~3 months post-treatment completion)
  Comparing institutional readmission as documented by CSC staff between treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: James MacKillop, PhD, CPsych, FCAHS, Principal Investigator — Peter Boris Centre for Addictions Research, St Joseph's Healthcare Hamilton
Locations (2):
- Canada (2):
  - The Salvation Army - Ellen Osler Home, Dundas, Ontario
  - The St. Leonard's Society Of Hamilton, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: No
Data from criminal justice-involved participants is considered sensitive and the Correctional Services of Canada prohibits the sharing of individual participant data with other organizations. Therefore, we will not be sharing IPD. Only aggregate and anonymized data in written research reports will be publicly shared.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-08): https://cdn.clinicaltrials.gov/large-docs/18/NCT07342218/Prot_SAP_000.pdf
  • Informed Consent Form (2025-09-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT07342218/ICF_001.pdf